CLINICAL TRIAL: NCT06309836
Title: Retrospective and Prospective Observational Study in Patients With Advanced Basal Cell Carcinoma
Acronym: REGISTRO-BCC
Status: Recruiting | Type: Observational
Sponsor: Societa Italiana di Dermatologia Medica, Chirurgica, Estetica e di Malattie Sessualmente Trasmesse (Other)
Responsible Party: Sponsor
Other Study IDs: SID03
Record Dates: First submitted 2023-08-04; First posted 2024-03-13 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Retrospective and Prospective Observational Study in Patients With Advanced Basal Cell Carcinoma.

DETAILED DESCRIPTION:
Basal cell carcinoma (BCC) is an epithelial tumor characterized by the malignant proliferation of keratinocytes in the basal layer of the epidermis. It is part, along with squamous cell carcinoma (SCC),non-melanoma skin cancer (NMSC) and accounts for 80% of all skin cancers and the most common skin cancer in the United States and Europe. Estimates of BCC incidence, however, are inaccurate since in most countries there is no cancer register collecting data on BCC incidence and many patients are treated on a territorial outpatient basis, making data collection and epidemiological analysis complex. In recent decades, there has been an increasing trend in patients with BCC, as well as a reduction in the average age of onset, with a consequent drastic increase in the social and economic cost of healthcare facilities. From these considerations, arises the need to investigate and characterize the profile of patients with advanced BCC, the clinical characteristics and the course of such neoplasm, and the choice of therapeutic options available.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged ≥ 18 years
2. Patients diagnosed with advanced basal cell carcinoma of the skin, i.e. tumours included in at least one of the following categories: locally advanced carcinoma (not radically treatable by surgery and/or radiotherapy), carcinoma with lymph node and/or distant metastatic localisation
3. patients who have had at least one access (first visit or follow-up visit) at the dermatology or oncology outpatient clinic of the centres involved

   * Patients diagnosed with advanced BCC who have accessed the centre from 1 January 2016 until the date of activation of the centre will be included in the retrospective cohort;
   * Patients diagnosed with advanced BCC who have accessed the centre from the date of activation
4. Signature of informed consent

Exclusion Criteria:

Patients incapable of giving informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with advanced basal cell carcinoma of the skin
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
clinical evolution, treatment and prognosis | from baseline through study completion, an average of 3 years
  clinical profile of patient, the phenotypic and behavioural characteristic and the clinical course from baseline to follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ketty MD Peris, Principal Investigator — IRCCS FONDAZIONE POLICLINICO GEMELLI
Locations (1):
- Irccs Fondazione Policlinico Gemelli, Roma, ITA, Italy